CLINICAL TRIAL: NCT06364865
Title: A Prospective, Observational Clinical Registry Study to Assess Safety and Performance of AE05ML Device for ML Hem-o-lok Polymer Clip Delivery in Laparoscopic Surgical Procedures
Brief Title: AE05ML Device for ML Hem-o-lok Polymer Clip Delivery in Laparoscopic Surgical Procedures Observational Registery Study
Acronym: AE05ML
Status: Enrolling by invitation | Type: Observational
Sponsor: Teleflex (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-04
Record Dates: First submitted 2024-04-02; First posted 2024-04-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Gall Bladder Disease; Bile Duct Diseases; Acute Cholecystitis; Kidney; Liver; Appendix; Spleen Disease; Prostate
MeSH Terms: conditions — Gallbladder Diseases; Bile Duct Diseases; Cholecystitis, Acute; Splenic Diseases | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: laparoscopic procedure — Not applicable, subject requiring procedure will have a laparoscopic procedure performed according to the institutions standard of care procedures. There are no clinical procedures performed on the subject as part of this registry study. Surgeon will answer questionnaires regarding use of the device upon completion of the laparoscopic procedure.

SUMMARY:
This clinical registry study aims to evaluate the safety and effectiveness of the AE05ML device for ligating vessels and tissue structures during laparoscopic surgery using Hem-o-lok® Medium Large (ML) polymer clips. The primary objective is to assess the device's safety and performance, with secondary objectives focusing on device performance characteristics and operator feedback.

DETAILED DESCRIPTION:
The objective of this clinical registry study is to evaluate safety and performance of the Weck® Auto Endo5® 5 mm automatic endoscopic 35 cm applier device (Teleflex Incorporated, Morrisville, NC, USA - further referred to as AE05ML) for delivery of Hem-o-lok® Medium Large (ML) polymer clips for the purpose of vessel / tissue structure ligation in laparoscopic surgery. This is a prospective, observational, multi-center, clinical registry study. All subjects will undergo vessel / tissue structure ligation using AE05ML during their indicated laparoscopic procedure as per standard of care and institutional policy and procedure.

The primary objective is to evaluate the safety and performance of AE05ML for delivery of ML Hem-o-lok polymer clips for the purpose of vessel / tissue structure ligation in adult subjects during laparoscopic procedures.

Primary Endpoints

* Safety: Incidence of device related adverse events (AE)
* Performance: Success / Failure of polymer clip delivery attempts The secondary objectives are to evaluate device performance characteristics and operator reported feedback regarding their experience using the device for each case.

Secondary Endpoint

• Results of Device Performance and Operator Feedback Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled for a laparoscopic procedure in which AE05ML will be used for vessel / tissue structure ligation
* Capable of providing informed consent for participation

Exclusion Criteria:

* Imprisoned
* Cognitively impaired and unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo laparoscopic procedures for which AE05ML is planned for use for delivery of ML Hem-o-lok polymer clips for ligation of vessels / tissue structures 3 - 10 mm in size, per the device instructions for use (IFU), should be considered for participation in the study. One hundred sixty-one (161) evaluable adult subjects are required. An evaluable subject is defined as a subject in whom clip delivery via AE05ML was attempted, during their scheduled laparoscopic procedure, in accordance with the device IFU, and the Laparoscopic Procedure Data Collection was performed. Additional subjects will be recruited to replace non-evaluable subjects to meet the target sample size. Reasons for determining a subject to be non-evaluable will be documented.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Evaluating the safety of AE05ML | Duration of AE05ML used during laparoscopic procedure
  The primary objective is to evaluate the safety (Incidence of device related adverse events (AE)) of AE05ML for delivery of ML Hem-o-lok polymer clips for the purpose of vessel / tissue structure ligation in adult subjects during laparoscopic procedures.
Evaluating the performance of AE05ML | Duration of AE05ML used during laparoscopic procedure
  The primary objective is to evaluate the performance (Success / Failure of polymer clip delivery attempts) of AE05ML for delivery of ML Hem-o-lok polymer clips for the purpose of vessel / tissue structure ligation in adult subjects during laparoscopic procedures.

SECONDARY OUTCOMES:
Evaluating device performance characteristics | Duration of AE05ML used during laparoscopic procedure
  The secondary objectives are to evaluate device performance characteristics of the AE05ML device during laparoscopic procedures by evaluating user reported feed back from user questionnaires.
Evaluating operator reported feedback | Duration of AE05ML used during laparoscopic procedure
  The secondary objectives are to evaluate operator reported feedback, on questionnaires, regarding their experience using the device for each case.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana A Puga, BS, Study Director — Teleflex Inc
Locations (3):
- United States (3):
  - Baptist Health South Miami, Miami, Florida
  - Northwell Health Long Island Jewish Hospital, New Hyde Park, New York
  - New Hanover Regional, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: No
Data will not be shared